CLINICAL TRIAL: NCT00266565
Title: A Phase I/II Study of the Effect of Intravenous Anti-IL-5 (Mepolizumab) SB 240563 on the Outcome and Management of Hypereosinophilic Syndromes
Brief Title: Anti-Interleukin-5 (IL-5) Study for Hypereosinophilic Syndrome
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 01-9-18; FD-R-002396 (Other: Cincinnati Childrens)
Record Dates: First submitted 2005-12-15; First posted 2005-12-19 (Estimated); Last update posted 2020-07-29 (Actual); Status verified 2020-07

CONDITIONS: Hypereosinophilic Syndromes; Eosinophilic Gastroenteritis; Churg-Strauss Syndrome; Eosinophilic Esophagitis
MeSH Terms: conditions — Hypereosinophilic Syndrome; Eosinophilic enteropathy; Churg-Strauss Syndrome; Eosinophilic Esophagitis | interventions — mepolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Anti-IL5 (Mepolizumab) (Experimental): The purpose of the study is to assess the toxicity of anti-IL-5 (Mepolizumab), and to see whether it lowers eosinophils in peripheral blood and/or tissue and whether it has a steroid and/or interferon sparing effect.
  Interventions: Drug: Mepolizumab

INTERVENTIONS:
Drug: Mepolizumab — 10mg/kg (max 750 ml) once a month for 3 months
  Other Names: Anti-IL5

SUMMARY:
Toxicity of anti-IL-5

DETAILED DESCRIPTION:
The purpose of the study is to assess the toxicity of anti-IL-5, and to see whether it lowers peripheral blood eosinophils and/or tissue and whether it has a steroid and/or interferon sparing effect.

ELIGIBILITY:
Inclusion Criteria:

* Adequate renal, cardiac, and hepatic function
* Not pregnant or breastfeeding
* A diagnosis of hypereosinophilic syndrome such as:

  * Idiopathic hypereosinophilic syndrome;
  * Eosinophilia myalgia syndrome;
  * Eosinophilic gastroenteritis;
  * Churg-Strauss syndrome;
  * Eosinophilic cellulitis;
  * Benign hypereosinophilia; or
  * Eosinophilic esophagitis.
* Maintained on, or in need of, the following: glucocorticoids, interferon, methotrexate, hydroxyurea, cytoxan, 6-mercaptopurine, or vincristine
* Blood eosinophil counts greater than 750 cells/mcl

Exclusion Criteria:

* Creatinine > 3 X upper limit for age
* AST > 5 X upper limit for age
* Platelet count < 50,000/mm3
* Cardiac function:

  1. NYHA class IIIb or IV (patients with shortness of breath or fatigue with mild exertion or at rest);
  2. Patients with symptomatic supraventricular or ventricular arrythmias requiring treatment;
  3. Patients requiring IV heart failure medications;
  4. Angina or acute myocardial infarction
* History of renal, hepatic, endocrine, oncologic, cardiovascular disease, or any other condition which, in the opinion of the Investigator, would jeopardize the safety of the patient or impact on the validity of the study results
* History of allergic or adverse response to previous antibody type therapy
* History of allergic or adverse response to anti-IL-5 therapy
* Evidence of, or history of, a parasitic infection (within past 1 year)
* Participation in a previous clinical trial involving an investigational agent within 30 days prior to study initiation
* Receipt of anti-IL-5 therapy in the past
* Blood donation of 450 ml (1 pint) or more within 30 days prior to study initiation
* Abnormal or unusual diet or substantial changes in eating habits within 30 days prior to, or during, the study.
* Patients who do not have eosinophil levels > 750 cells/mcl after the run-in period. Patients who have only eosinophilic infiltration of tissue are eligible if they do not develop an eosinophil level > 750 cells/mcl, assuming that they meet all other eligibility requirements.
* Positive serum pregnancy test
* Breastfeeding
* Unable to use effective birth control methods for duration of study
* Unable or unwilling to give voluntary informed consent/assent

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2001-12 (Actual); Primary Completion 2005-04 (Actual); Study Completion 2005-04 (Actual)

PRIMARY OUTCOMES:
To assess the toxicity of anti-IL-5 in patients with hypereosinophilia | 28 weeks

SECONDARY OUTCOMES:
To assess whether anti-IL-5 lowers peripheral blood eosinophils and/or tissue in patients with hypereosinophilia | 28 weeks
To assess whether anti-IL-5 has a steroid and/or interferon sparing effect | 28 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Marc E. Rothenberg, MD, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States